CLINICAL TRIAL: NCT02441543
Title: Regulation of Lymphocyte Anti-tumor Response in Metastatic Patients Treated With the mTOR Inhibitor Everolimus
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: ONC/OSS-01/2015
Record Dates: First submitted 2015-04-28; First posted 2015-05-12 (Estimated); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: SOLID TUMOR

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No

SUMMARY:
Preclinical studies and clinical observations have shown the Phosphoinositide 3-kinase (PI3K) /Protein kinase B (AKT) /mammalian (mechanistic) target of Rapamycin (known as the 'mTOR-pathway') signaling to be deregulated in several tumors.

DETAILED DESCRIPTION:
Cancer is the second most-common cause of death in industrialized countries. Preclinical studies and clinical observations have shown the PI3K/AKT/mammalian (mechanistic) target of Rapamycin (known as the 'mTOR-pathway') signaling to be deregulated in several tumors.

The mTOR is evolutionary conserved Serine/Threonine protein kinase that senses and integrates signals from different environmental cues. It is a central regulator of cell growth, cell cycle progression, proliferation and metabolism. It has been found to form two distinct, multiprotein complexes based on the binding with different partners. In a complex with Regulatory-Associated Protein of mTOR (Raptor) mTOR forms mTORC1, whereas when bound to Rapamycin-Insensitive Companion of mTOR (Rictor) than the mTOR Complex 2 (mTORC2) is formed. Not only the structure of both mTOR complexes is different, but also they are characterized by distinct biological functions mediated by individual downstream targets. The mTORC1 promotes cap-dependent translation and elongation, increases Messenger RNA (mRNA) biogenesis as well as promotes ribosome biogenesis - via regulation of p70 ribosomal S6 kinase 1 (p70S6K) as well as the eukaryotic initiation factor 4E (eIF4E) binding protein 1 (4EBP-1). In addition mTORC1 promotes lipid synthesis via sterol regulatory element binding protein 1 (SREBP1) and peroxisome proliferator-activated receptor-γ (PPARγ). The role of the mTORC2 is less defined. The best characterized, mTORC2 target is AKT, which regulates cell survival, metabolism and proliferation as well as differentiation in many primary and cancer cell types. Another direct targets of mTORC2 are the serum- and glucocorticoid-regulated kinase (SGK) controls cell survival and anabolism and protein kinase Cα (PKCα) involved in the control of cytoskeletal organization. Thus constitutive, oncogenic activation of mTOR signaling promotes protein and lipid synthesis needed for the increase in cell mass and it enhances surface transporters expression sustaining better uptake of glucose, amino acids and other nutrients sustaining cell growth and proliferation of transformed cells.

Since mTOR signalling pathway is critical for tumorigenesis, its inhibitors have been strongly wanted. As first approved by FDA in clinical setting was Rapamycin for its activity against transplant organ rejection and as a prophylactic agent in Graft-versus-Host disease after allogenic bone marrow transplantation. The immunosuppressive effects of Rapamycin were initially attributed to its ability to block the Interleukin 2 (IL-2) induced proliferation. However, later this was found not to be the case, and rather work through immunomodulation, in part due to the induction and expansion of T cells with regulatory phenotype. Moreover, in T cells mTORC1 modulates T helper cell differentiation towards Th1 and Th17 fate, while mTORC2 controls Th2 development. Also, Rapamycin is involved in immunostimulation of long-lived memory cluster of differentiation 8+ (CD8+) T cells. In addition to the Rapamycin effect on T cells, the drug exerts an inhibitory effect on the proliferation and function of other immune cells such as dendritic cells, B lymphocytes, Natural Killer cells (NK), neutrophiles and mast cells. Lastly, Rapamycin has been tested as a chemotherapy agent against cancer and it was shown to delay the growth and proliferation and to promote apoptosis of many cancer cell lines, and also to possess anti-angiogenic properties. During the past years different rapalogs have been synthesized among which is Everolimus (RAD001, Afinitor®) that is currently tested in clinical trials phase IV in patients with renal cell carcinoma (RCC) or advance large cell lung cancer with neuroendocrine differentiation as well as in the phase III of metastatic breast cancer. In addition, it is already approved in different tumors when the first-line treatment was ineffective. Even Everolimus seems to be very promising neoplastic agent, there is no clinical data about its effect on the immune competence of the patients. And it still remains unknown whether Everolimus exerts similar to Rapamycin effect on the modulation of the immune system when administrated into cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic tumor cancer
* Treated with Everolimus

Exclusion Criteria:

* Non metastatic tumor
* Non previously treated with Everolimus

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Metastatic tumor patients treated with Everolimus
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2015-04; Primary Completion 2018-04 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Sensitivity of mTORC1 and mTORC2 | 3 years
  Evaluate the sensitivity of mTORC1 and mTORC2 to Everolimus in T and NK cells.Everolimus inhibits kinase activity of mTOR when bound to Raptor (mTORC1). Whether mTORC2 is sensitive to Everolimus will be elucidated.

SECONDARY OUTCOMES:
Determine the phenotype of T cells. | 3 years
  Determine the phenotype of T cells in patients with the use of mass cytometry and polychromatic flow cytometry. Everolimus alters the phenotype and dynamics of circulating T and NK cells.
Evaluate the ability of T-cells | 3 years
  Evaluate the ability of T-cells from patients to differentiate into effector cells (anti-tumor and anti- viral in vitro responses. Everolimus potentiates anti-tumor and anti-viral immune responses and that will affect the differentiation of naive T cell precursors into memory cells

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Lugli, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- Istituto Clinico Humanitas, Rozzano, MI, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zoncu R, Efeyan A, Sabatini DM. mTOR: from growth signal integration to cancer, diabetes and ageing. Nat Rev Mol Cell Biol. 2011 Jan;12(1):21-35. doi: 10.1038/nrm3025. Epub 2010 Dec 15. PMID 21157483
- [Background] Battaglia M, Stabilini A, Roncarolo MG. Rapamycin selectively expands CD4+CD25+FoxP3+ regulatory T cells. Blood. 2005 Jun 15;105(12):4743-8. doi: 10.1182/blood-2004-10-3932. Epub 2005 Mar 3. PMID 15746082
- [Background] Powell JD, Pollizzi KN, Heikamp EB, Horton MR. Regulation of immune responses by mTOR. Annu Rev Immunol. 2012;30:39-68. doi: 10.1146/annurev-immunol-020711-075024. Epub 2011 Nov 29. PMID 22136167
- [Background] Hasskarl J. Everolimus. Recent Results Cancer Res. 2014;201:373-92. doi: 10.1007/978-3-642-54490-3_23. PMID 24756805
- [Background] Zeng Z, Sarbassov dos D, Samudio IJ, Yee KW, Munsell MF, Ellen Jackson C, Giles FJ, Sabatini DM, Andreeff M, Konopleva M. Rapamycin derivatives reduce mTORC2 signaling and inhibit AKT activation in AML. Blood. 2007 Apr 15;109(8):3509-12. doi: 10.1182/blood-2006-06-030833. Epub 2006 Dec 19. PMID 17179228
- [Background] Bachelot T, Bourgier C, Cropet C, Ray-Coquard I, Ferrero JM, Freyer G, Abadie-Lacourtoisie S, Eymard JC, Debled M, Spaeth D, Legouffe E, Allouache D, El Kouri C, Pujade-Lauraine E. Randomized phase II trial of everolimus in combination with tamoxifen in patients with hormone receptor-positive, human epidermal growth factor receptor 2-negative metastatic breast cancer with prior exposure to aromatase inhibitors: a GINECO study. J Clin Oncol. 2012 Aug 1;30(22):2718-24. doi: 10.1200/JCO.2011.39.0708. Epub 2012 May 7. PMID 22565002
- [Background] Bendall SC, Simonds EF, Qiu P, Amir el-AD, Krutzik PO, Finck R, Bruggner RV, Melamed R, Trejo A, Ornatsky OI, Balderas RS, Plevritis SK, Sachs K, Pe'er D, Tanner SD, Nolan GP. Single-cell mass cytometry of differential immune and drug responses across a human hematopoietic continuum. Science. 2011 May 6;332(6030):687-96. doi: 10.1126/science.1198704. PMID 21551058
- [Background] Lugli E, Gattinoni L, Roberto A, Mavilio D, Price DA, Restifo NP, Roederer M. Identification, isolation and in vitro expansion of human and nonhuman primate T stem cell memory cells. Nat Protoc. 2013 Jan;8(1):33-42. doi: 10.1038/nprot.2012.143. Epub 2012 Dec 6. PMID 23222456
- [Background] Motzer RJ, Escudier B, Oudard S, Hutson TE, Porta C, Bracarda S, Grunwald V, Thompson JA, Figlin RA, Hollaender N, Kay A, Ravaud A; RECORD-1 Study Group. Phase 3 trial of everolimus for metastatic renal cell carcinoma : final results and analysis of prognostic factors. Cancer. 2010 Sep 15;116(18):4256-65. doi: 10.1002/cncr.25219. PMID 20549832
- [Background] Cieri N, Camisa B, Cocchiarella F, Forcato M, Oliveira G, Provasi E, Bondanza A, Bordignon C, Peccatori J, Ciceri F, Lupo-Stanghellini MT, Mavilio F, Mondino A, Bicciato S, Recchia A, Bonini C. IL-7 and IL-15 instruct the generation of human memory stem T cells from naive precursors. Blood. 2013 Jan 24;121(4):573-84. doi: 10.1182/blood-2012-05-431718. Epub 2012 Nov 15. PMID 23160470